CLINICAL TRIAL: NCT05492955
Title: Implementation of a Combination Intervention for Sustainable Blood Pressure Control in KwaZulu-Natal, South Africa (IMPACT-BP)
Brief Title: Implementation of a Combination Intervention for Sustainable Blood Pressure Control
Acronym: IMPACT-BP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Thomas A Gaziano, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021P003469
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard of Care (SOC) (Active Comparator): Participants will receive clinic-based standard of care
  Interventions: Behavioral: Standard of Care Model
- Community Health Worker Care Model (CHW) (Experimental): Participants will be given a standard blood pressure cuff (Omron) for at-home BP monitoring, and will be assigned to a CHW for follow-up visits and medication delivery.
  Interventions: Behavioral: Community Health Worker Care Model
- Enhanced Community Health Worker + Mobile Health Monitoring (eCHW+) (Experimental): Participants will be given a blood pressure cuff with cellular capability (Blipcare) for at-home BP monitoring which automatically transmit BP data to our server for nurse review. These participants will also be assigned to a CHW for follow-up visits and medication delivery.
  Interventions: Behavioral: Enhanced Community Health Worker-based with Mobile Health Blood Pressure Monitoring Model

INTERVENTIONS:
Behavioral: Community Health Worker Care Model — Participants will be given a digital BP Cuff and a standardized training on its operation, and assigned a CHW from their local Community Health Team. The participant will be instructed to take 6-10 measurements BP per week and record them in a logbook. CHWs will return to participant homes every 2-4 weeks to collect BP measurements and enter them into a data collection system, assess for symptoms, and discuss treatment adherence and lifestyle recommendations. BP readings will be brought by the CHW to their assigned nursing supervisors at their local clinic, who will initiate and tailor medications based on a standardized clinical decision support algorithm, based on SA DoH hypertension control guidelines. All treatment decisions will be made by the nursing supervisors. Participants will either obtain medication(s) at the pharmacy or, as possible, have them delivered by a CHW.
  Other Names: CHW Model
  Arms: Community Health Worker Care Model (CHW)
Behavioral: Enhanced Community Health Worker-based with Mobile Health Blood Pressure Monitoring Model — Participants in this arm will also be given a BP Cuff, (but with cellular network capability, such that BP data can be directly transmitted to trial server), given training on its operation, and assigned a CHW from their local Community Health Team. The participant will be instructed to take 6-10 measurements BP per week, which will be automatically uploaded onto the server to be made available by the nurse supervisors. CHWs will return to participant homes every 2-4 weeks to ensure functionality of the devices and transmission, collect BP measurements if the system is not functional, assess for symptoms, and discuss treatment adherence and lifestyle recommendations. Nursing supervisors at the clinic will use the remotely collected BP data to initiate and tailor medications based on the same standardized clinical decision support (CDS) algorithm, based on SA DoH hypertension control guidelines. All treatment decisions will be made by the nursing supervisors.
  Other Names: eCHW+ Model
  Arms: Enhanced Community Health Worker + Mobile Health Monitoring (eCHW+)
Behavioral: Standard of Care Model — Participants in the SOC arm will be referred to their clinic for active care as per standard clinical protocols. All care will be provided at the clinic. Routine care consists of regular visits to the clinic until BP is under control (<140/90 mmHg) and then at 6 monthly intervals. BP measurements to guide management decisions will be made at the clinic using standard clinic equipment. Symptoms related to hypertension and/or medications will be assessed at each visit. Medications available will include medications on the South African Essential Drug list and which are available in the pharmacy. Prescriptions are picked up at the clinic pharmacy by patients as per routine protocol at the clinics. CHWs may also conduct monitoring as guided by clinical guidelines and as advised by their clinical supervisors during the study period to assess for adherence and provide education.
  Other Names: SOC Model
  Arms: Standard of Care (SOC)

SUMMARY:
This is a randomized clinical trial intended to identify the optimal strategy of blood pressure management in rural South Africa using Community Health Workers (CHWs) in conjunction with in-home BP monitoring among adults.

DETAILED DESCRIPTION:
We will conduct a trial using CHWs in conjunction with in-home BP monitoring among 774 adults ≥ 18 years old residing in uMkhanyakude District in northern KwaZulu-Natal in an area that is served by a CHW. Eligible participants will be recruited from prior community-based hypertension screening programs, CHW-led hypertension screening activities, and/or from trial clinics where they are accessing care. Consenting participants will be randomized to one of the three study arms of hypertension care (258 participants per arm): 1) clinic-based standard of care model (SOC); 2) community health worker-based blood pressure monitoring model (CHW); 3) and enhanced community health worker-based model, including mobile health blood pressure monitoring model (eCHW+). Independent of clinical care, all participants will be seen at enrollment and at 6 months for BP monitoring and data collection by study nurses for outcome assessments. The primary effectiveness outcome will be assessed in an intention-to-treat analysis and defined as the change in systolic blood pressure (SBP) 6 months after enrollment. The secondary effectiveness outcome will be the proportion of participants with controlled blood pressure, as defined by an SBP <140 mmHg and a diastolic BP (DBP) <90 mmHg 6 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years old
* Residing in uMkhanyakude District in northern KwaZulu-Natal in an area that is served by a CHW.
* Elevated blood pressure (blood pressure > 140/90 mmHg) on two measurements.

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Severe, symptomatic hypertension with a measured blood pressure > 180/110 mmHg.
* Known, advanced chronic kidney disease. GFR < 60 ml/min/1.73 m2.
* Current use of at least 3 different anti-hypertensive therapies at full dose.
* Planning to move within the next 24 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 774 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
Mean systolic blood pressure change | 6 months
  Absolute change in systolic blood pressure (SBP) between baseline and 6 months after enrollment.

SECONDARY OUTCOMES:
Achievement of blood pressure control | 6 months
  Blood pressure control, defined as a BP <140/90 6 months after enrollment

OTHER OUTCOMES:
Adverse events (safety) | 6 months
  Number of adverse and severe adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Gaziano, MD, MSc, Principal Investigator — Massachusetts General Hospital; Mark J Siedner, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Africa Health Research Institute (AHRI), Mtubatuba, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the study, in compliance with guidance by the study funders (U.S. National Institutes of Health), study data will be fully de-identified and posted to a public data repository where it may be shared with other scientists for secondary use.
Supporting Information: Study Protocol, ICF
Time Frame: After completion of study, data cleaning, and prespecified analyses.
Access Criteria: Because of the sensitive nature of the data collected for this study, requests to access the data set from qualiﬁed researchers trained in human subject conﬁdentiality protocols may be sent to the primary investigator.

REFERENCES:
- [Derived] Siedner MJ, Magula N, Mazibuko L, Sithole N, Castle A, Nxumalo S, Manyaapelo T, Abrahams-Gessel S, Gareta D, Orne-Gliemann J, Baisley K, Bachmann M, Gaziano TA. Home-Based Care for Hypertension in Rural South Africa. N Engl J Med. 2025 Oct 2;393(13):1304-1314. doi: 10.1056/NEJMoa2509958. Epub 2025 Sep 1. PMID 40888742